CLINICAL TRIAL: NCT01211977
Title: A Pilot Study of XOMA 052 in Familial Cold Autoinflammatory Syndrome (FCAS) / Muckle-Wells Syndrome (MWS) and Behcet's Disease (BD)
Brief Title: A Pilot Study of XOMA 052 in Familial Cold Autoinflammatory Syndrome / Muckle-Wells Syndrome and Behcet's Disease
Status: Withdrawn | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: National Institute of Arthritis and Musculoskeletal and Skin Diseases (NIAMS) (NIH)
Responsible Party: Cailin C. Henderson, M.D./National Institute of Arthritis and Musculoskeletal and Skin Diseases, National Institutes of Health
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: 100182; 10-AR-0182
Record Dates: First submitted 2010-09-29; First posted 2010-09-30 (Estimated); Last update posted 2017-07-02 (Actual); Status verified 2011-04-29

CONDITIONS: Muckle Wells Syndrome; Autoinflammatory; Behcet's Disease
Keywords: Muckle Wells Syndrome; Autoinflammatory; Interleukin-1
MeSH Terms: conditions — Cryopyrin-Associated Periodic Syndromes; Behcet Syndrome | interventions — gevokizumab

INTERVENTIONS:
Drug: XOMA 052

SUMMARY:
Background:

* Autoinflammatory diseases are illnesses that produce episodes of inflammation such as fever, rash, or joint swelling. Some of these diseases can be treated with medications that block the body's reaction to a protein called IL-1, which may be part of the cause of the inflammation. IL-1 blocking agents are very helpful in treating autoinflammatory diseases and have become the standard of care for treatment for some of these diseases. However, more research is needed on related diseases that may be treated with new and currently used IL-1 blocking agents.
* XOMA 052 is an experimental drug that is currently being tested as a possible treatment for type 2 diabetes. Initial studies have shown that XOMA 052 neutralizes a specific kind of IL-1, and is also active against certain indicators of inflammation. Researchers are interested in determining whether XOMA 052 can be used to treat autoinflammatory and related diseases.

Objectives:

- To determine the effectiveness of XOMA 052 as a treatment for inflammation in adults with the autoinflammatory diseases Familial Cold Autoinflammatory Syndrome (FCAS)/Muckle-Wells Syndrome (MWS) and Behcet's Disease.

Eligibility:

* FCAS/ MWS: Individuals at least 18 years of age who have a known history of the typical disease.
* Behcet's Disease: Individuals at least 18 years of age who have evidence of active disease, such as oral or genital ulcers or eye disease.

Design:

FCAS/MWS Participants

* Participants will have an overnight evaluation of their disease, including optional tests (e.g., eye or skin exams). Participants who currently take medications to treat their symptoms will stop taking the medication and will be monitored by study researchers. At the first flare of symptoms, participants will begin to receive XOMA 052.
* Participants will have further tests on days 3, 7, and 10 after the initial dose of XOMA 052. If the disease remains under good control, participants will have a clinical exam every 5 days for up to 10 weeks until another disease flare occurs (determined either by symptoms or by inflammation observed in laboratory studies). If the disease is not well controlled with the initial dose of XOMA 052, participants will have additional doses starting at day 7 until either the disease is controlled or researchers determine that the medication is not effective.
* Participants will have the option to continue XOMA 052 treatments for up to 1 year. XOMA 052 wil...

DETAILED DESCRIPTION:
Autoinflammatory diseases are illnesses characterized by episodes of inflammation that, unlike autoimmune disorders, lack the production of high titer autoantibodies or antigen-specific T cells. There is growing genetic and clinical evidence that Interleukin-1 (IL-1) plays a pathogenic role in several of these diseases. This exploratory study aims to examine the utility of the experimental drug candidate, XOMA 052 (XOMA (US), LLC) in the treatment of adult subjects with the autoinflammatory disorders familial cold autoinflammatory syndrome (FCAS) or Muckle-Wells Syndrome (MWS) associated with mutations in cryopyrin-encoding CIAS1 and in adult subjects with Behcet's Disease (BD), a disease which may be responsive to IL-1 blockade. XOMA 052 is a human recombinant IL-1beta antibody with picomolar affinity for IL-1beta and a beta half-life of 22.4 days in humans. This agent is currently in Phase 2 clinical studies for the treatment of Type 2 Diabetes and initial studies have shown activity against clinical and biochemical indicators of inflammation.

This pilot study is designed to address: 1) the utility of XOMA 052 in the treatment of FCAS / MWS, in a disease known to respond to IL-1 blockade (FCAS / MWS) as shown by a response to treatment with anakinra (Kineret(Registered Trademark), recombinant IL-1 receptor antagonist), rilonacept (Arcalyst(Registered Trademark), IL-1 Trap, a fusion protein of the IL-1 receptor and the Fc portion of IgG), and canakinumab (Ilaris(Registered Trademark), IL-1beta blocking antibody); the latter two FDA approved for the treatment of this condition; 2) the pharmacokinetics and dynamics of treatment with XOMA 052 in FCAS / MWS; 3) the effect of XOMA 052 on laboratory biomarkers in BD; and 4) an exploratory assessment of the utility of XOMA 052 in the treatment of BD.

For FCAS / MWS, biochemical and clinical correlates of autoinflammatory disease will be measured at baseline following withdrawal of currently used IL-1 inhibitors. Subjects will receive a course of therapy with XOMA 052 that is predicted to provide an estimated 4 weeks of anti-inflammatory activity. If a favorable response is obtained, the continuation phase will last twelve months. For BD, subjects will receive XOMA 052 for three to six months and patients with a positive response will then be randomized to withdrawal or continuation of drug for six months. Clinical and biochemical correlates of inflammation will be measured in both patient groups at appropriate intervals to assess response and to further elucidate disease mechanisms.

ELIGIBILITY:
* INCLUSION CRITERIA:

FOR FCAS / MWS:

1. Male or female subjects with inflammatory disease greater than or equal to 18 years of age.
2. Participation in NIH study #03-AR-0173 ( Studies of the Natural History, Pathogenesis, and Outcome of Autoinflammatory Diseases )
3. CIAS1 mutation positivity or FCAS / MWS based on clinical grounds with a history of a complete response to IL-1 blocking medications.
4. Subjects presenting with active FCAS / MWS based on clinical signs/symptoms in addition to elevated acute phase reactants (CRP, SAA or ESR). To meet established clinical criteria for active disease, patients must have recurrent intermittent episodes of fever and rash, an age of onset < 6 months of age, duration of most attacks < 24 hours, and the presence of conjunctivitis with attacks. Active disease will be defined as either the presence of classical features or a history of such features that became quiescent in the setting of therapy with anakinra or rilonacept. However, before a patient who has quiescent disease and is currently taking anakinra or rilonacept can receive study drug, he/she must fulfill criteria for active disease after anakinra or rilonacept has been discontinued. Subjects must be greater than 48 hours from their last dose of anakinra (half-life 4-6 hours) and 14 days from their last dose of rilonacept (half-life 7.5 days) before beginning XOMA 052 therapy, and will not take anakinra or rilonacept for the remainder of their enrollment in the study.
5. Stable dose of steroids, NSAIDs, DMARDs, or colchicine for four weeks prior to enrollment visit.
6. Females of childbearing potential (young women who have had at least one menstrual period regardless of age) must have a negative urine pregnancy test at screening and a negative serum pregnancy test at baseline prior to performance of any radiologic procedure or administration of study medication.
7. Women of childbearing age and men able to father a child, who are sexually active, who agree to use a form of effective birth control, including abstinence.
8. Either (1) a negative PPD test using 5 T.U. intradermal testing per CDC guidelines and no evidence of active TB by history on chest X-ray at the time of enrollment or (2) a positive PPD with no evidence of active TB on chest X-ray at the time of enrollment and either past or present treatment with adequate therapy for at least one month prior to first dose of study medication. Full prophylaxis regimens will be completed. Subjects who have been BCG-vaccinated will also be skin-tested.
9. Able to understand, and complete study-related questionnaires.
10. Able and willing to give informed consent and abide with the study procedures.

FOR BD:

1. Male or female subjects with BD associated inflammatory disease greater than or equal to 18 years of age.
2. Participation in NIH study #03-AR-0173 ( Studies of the Natural History, Pathogenesis, and Outcome of Autoinflammatory Diseases )
3. Diagnosis of Behcet's disease as determined by the International Study Group Criteria or by complete Japanese Criteria
4. Active mucocutaneous disease as defined by at least one oral or genital ulcer within the past month.
5. Stable dose of steroids, NSAIDs, DMARDs, or colchicine for four weeks prior to enrollment visit.
6. For patients with ocular disease, no active intermediate or posterior disease at enrolment but history of an ocular flare (greater than or equal to 3 in the last 6 months) in the presence of any systemic anti-inflammatory therapy such as prednisone, azathioprine, Mycophenolate, methotrexate, cyclosporine, a TNF inhibitor, or a combination of these medications. Patients must have developed active disease in the presence of at treatment with at least one of the following medications for at least six months: azathioprine, cyclosporine, or a TNF inhibitor.
7. Females of childbearing potential (young women who have had at least one menstrual period regardless of age) must have a negative urine pregnancy test at screening and a negative serum pregnancy test at baseline prior to performance of any radiologic procedure or administration of study medication. Female patients will be screened for pregnancy at all NIH visits.
8. Women of childbearing age and men able to father a child, who are sexually active, who agree to use a form of effective birth control, including abstinence.
9. Either (1) a negative PPD test using 5 T.U. intradermal testing per CDC guidelines and no evidence of active TB on chest X-ray at the time of enrollment or (2) a positive PPD with no evidence of active TB by history or on chest X-ray at the time of enrollment and either past or present treatment with adequate therapy for at least one month prior to first dose of study medication. Full prophylaxis regimens will be completed. Subjects who have been BCG-vaccinated will also be skin-tested.
10. Able to understand, and complete study-related questionnaires.
11. Able and willing to give informed consent and abide with the study procedures.

EXCLUSION CRITERIA:

For both study populations:

1. Treatment with a live virus vaccine during 3 months prior to baseline visit. No live vaccines will be allowed throughout the course of this study.
2. Patients with ocular disease who received local treatments other than eye drops (i.e. periocular or intraocular steroids, implants or other antinflammatory agents within 4 weeks prior to enrollment)
3. Current treatment with TNF inhibitors or discontinuation of TNF inhibitors within 8 weeks.
4. Presence of active infections or a history of pulmonary TB infection with or without documented adequate therapy.
5. Chest x-ray read by a radiologist with pleural scarring and/or calcified granuloma consistent with prior TB.
6. Positive test for or prior history of HIV, Hepatitis B or C.
7. History or concomitant diagnosis of congestive heart failure.
8. History of malignancy. Subjects deemed cured of superficial malignancies such as cutaneous basal or squamous cell carcinomas, or in situ cervical cancer may be enrolled.
9. Known hypersensitivity to CHO cell derived biologicals or any components of XOMA 052.
10. Presence of any additional rheumatic disease or significant systemic disease. For example, major chronic infectious/ inflammatory/ immunologic disease (such as inflammatory bowel disease, psoriatic arthritis, spondyloarthropathy, SLE in addition to autoinflammatory disease).
11. Presence of any of the following laboratory abnormalities at enrollment visit: creatinine> 1.5 times the ULN, WBC< 3.6x10(9)/mm(3); platelet count < 75,000 mm(3); ALT or AST > 2.0 times the ULN
12. Lactating females or pregnant females.
13. Subjects with asthma not adequately controlled on current inhaled therapy for at least four weeks.
14. Enrollment in any other investigational treatment study or use of an investigational agent, or has not yet completed at least 4 weeks or 5 half-lives, whichever is longer, since ending another investigational device or drug trial.
15. Subjects for whom there is concern about compliance with the protocol procedures.
16. Presence of other severe acute or chronic medical or psychiatric condition, or significant laboratory abnormality requiring further investigation that may cause undue risk for the subject's safety, inhibit protocol participation, or interfere with interpretation of study results, and in the judgment of the investigator would make the subject inappropriate for entry into this study.
17. Treatment within the past 12 months with canakinumab
18. Active neurologic disease which would require cyclophosphamide treatment. Active neurologic disease is defined as either new evidence of parenchymal (meningoencephalitis) or non-parenchymal (vascular complications including thrombosis) disease.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2010-08-27; Primary Completion 2011-04-29 (Actual); Study Completion 2011-04-29 (Actual)

PRIMARY OUTCOMES:
Changes in clinical and biochemical indicators of inflammation
Safety

SECONDARY OUTCOMES:
Duration of response to single dose
Long term clinical and biochemical responses
Number of flares during randomized withdrawal
If applicable, assessment of the lack of complete response in relation to pharmacologic parameters.

CONTACTS AND LOCATIONS:
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Aksentijevich I, Putnam CD, Remmers EF, Mueller JL, Le J, Kolodner RD, Moak Z, Chuang M, Austin F, Goldbach-Mansky R, Hoffman HM, Kastner DL. The clinical continuum of cryopyrinopathies: novel CIAS1 mutations in North American patients and a new cryopyrin model. Arthritis Rheum. 2007 Apr;56(4):1273-1285. doi: 10.1002/art.22491. PMID 17393462
- [Background] Aksentijevich I, Nowak M, Mallah M, Chae JJ, Watford WT, Hofmann SR, Stein L, Russo R, Goldsmith D, Dent P, Rosenberg HF, Austin F, Remmers EF, Balow JE Jr, Rosenzweig S, Komarow H, Shoham NG, Wood G, Jones J, Mangra N, Carrero H, Adams BS, Moore TL, Schikler K, Hoffman H, Lovell DJ, Lipnick R, Barron K, O'Shea JJ, Kastner DL, Goldbach-Mansky R. De novo CIAS1 mutations, cytokine activation, and evidence for genetic heterogeneity in patients with neonatal-onset multisystem inflammatory disease (NOMID): a new member of the expanding family of pyrin-associated autoinflammatory diseases. Arthritis Rheum. 2002 Dec;46(12):3340-8. doi: 10.1002/art.10688. PMID 12483741
- [Background] Feldmann J, Prieur AM, Quartier P, Berquin P, Certain S, Cortis E, Teillac-Hamel D, Fischer A, de Saint Basile G. Chronic infantile neurological cutaneous and articular syndrome is caused by mutations in CIAS1, a gene highly expressed in polymorphonuclear cells and chondrocytes. Am J Hum Genet. 2002 Jul;71(1):198-203. doi: 10.1086/341357. Epub 2002 May 24. PMID 12032915